CLINICAL TRIAL: NCT05094700
Title: A Single Center, Monadic, Open Label, Four-Week Clinical Trial to Evaluate the Tolerance and of a Polymeric Surfactant Technology Cleanser in Sensitive Skin Patients
Brief Title: A Study of a Polymeric Surfactant Technology Cleanser in Sensitive Skin Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCSSKA004090; CCSSKA004090 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Dermatitis, Atopic; Rosacea; Acne Vulgaris; Sensitive Skin
MeSH Terms: conditions — Dermatitis, Atopic; Rosacea; Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-marketed Cosmetic Facial Cleanser (Experimental): Participants will receive non-marketed cosmetic facial cleanser to apply on cleanse facial skin, twice daily for 4 weeks.
  Interventions: Other: Non-marketed Cosmetic Facial Cleanser

INTERVENTIONS:
Other: Non-marketed Cosmetic Facial Cleanser — Participants will apply non-marketed cosmetic facial cleanser on cleanse facial skin, twice daily for 4 weeks.

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerance of a gentle facial cleanser in participants with sensitive skin (eczema/atopic dermatitis, rosacea, acne, cosmetic intolerance syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-70 years of age. Participants who are over 65 years of age must be Coronavirus Disease 2019 (COVID-19) vaccinated. The site will review state issued vaccination cards as proof of vaccination
* Fitzpatrick Skin Type I-VI, across a range of races and ethnicities with at least 2 participants per each Fitzpatrick skin type
* Participants who possess mild to moderate eczema/atopic dermatitis, mild to moderate rosacea, mild to moderate acne, or mild to moderate cosmetic intolerance syndrome
* Participants willing to continue normal course of treatment (within the past 30 days) for their skin disease/condition with no changes during the study
* Participants must provide written informed consent including consent for photograph release including Health Insurance Portability and Accountability Act (HIPAA) disclosure
* Able to read, write, speak, and understand English
* Generally in good health based on medical history reported by the participant
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

* Has very sensitive skin and/or has known allergies or adverse reactions to common topical skincare products or to ingredients in the investigational product (IP) or have demonstrated a previous hypersensitivity reaction to any of the ingredients in the IP
* Participants who are pregnant, breast feeding, or planning to become pregnant
* Participants with clinically significant unstable medical disorders
* Participants who are unwilling or unable to comply with the requirements of the protocol
* Participants who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study
* Participants with any planned surgeries and/or invasive medical procedures during the course of the study
* Participants who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study
* Presents with a skin or condition that, in the principal investigator (PI) or designee's opinion, may confound the study results or otherwise be inappropriate for study participation (example, pre-existing or dormant facial dermatologic conditions specifically severe acne or acne conglobata, psoriasis, rosacea, rashes, eczema, atopic dermatitis, skin cancer, many and/or severe excoriations, observable suntan, scars, nevi, tattoo, excessive hair, Et cetera [etc])
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including: a) Immunosuppressive or steroidal drugs within 2 months before Visit 1; b) Non-steroidal anti-inflammatory drugs within 5 days before Visit 1; c) Antihistamines within 2 weeks before Visit 1
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Is simultaneously participating in any other product-use study or has participated in another clinical study on the face in the past 4 weeks
* Participants currently receiving any anticancer, immunosuppressive treatments/medications (example, azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.), or radiation as determined by study documentation
* Participants with a history of immunosuppression/immune deficiency disorders (including [human immunodeficiency virus {HIV} infection or acquired immunodeficiency syndrome {AIDS})
* Is participating or receiving any professional or aesthetic facial spa procedures during the study
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor
* Has a history of a confirmed COVID-19 infection within 30 days prior to Visit 1
* Has had contact with a COVID-19-infected person within 14 days prior to Visit 1
* Individual or a member of the individual's household has traveled internationally within 14 days prior to Visit 1
* Has experienced any of the following self-reported symptoms of COVID-19 within 2 weeks prior to Visit 1: a) Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomachaches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever, or chest pain/tightness; b) Temperature greater than or equal to (>=) 37.5 degree Celsius (°C) / 99.5 degree Fahrenheit (°F), measured; c) Use of fever reducers within 2 days prior to each on-site visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Mildness of the Facial Cleanser in Participants with Sensitive Skin Based on Investigator and Participant Assessments | Baseline to Week 4
  Mildness of the facial cleanser in participants with sensitive skin (eczema/atopic dermatitis, rosacea, acne, cosmetic intolerance syndrome) based on investigator and participant assessments will be reported. It will be evaluated on a scale of 0 to 4 with 0=none, 1=almost clear, 2=mild, 3=moderate, 4=severe.

SECONDARY OUTCOMES:
Investigator Assessment for Tolerability | Baseline, Week 2 and Week 4
  Investigator observed tolerability parameters such as: redness/erythema, rash/irritation, peeling/flaking, tactile roughness, and dryness which will be measured using a 5-point ordinal scale (0=none, 1=minimal, 2=mild, 3=moderate, 4=severe).
Investigator Assessment for Efficacy | Baseline, Week 2 and Week 4
  Investigators observed efficacy parameters such as: visual smoothness, tactile softness, clarity, radiance, pores, and overall skin appearance which will be measured using a 5-point ordinal scale (0=none, 1=minimal, 2=mild, 3=moderate, 4=severe).
Participant Assessment for Tolerability | Baseline, Week 2 and Week 4
  Participants observed tolerability parameters such as: stinging, burning, itching, tightness, redness, flaking/peeling, roughness, dryness and overall sensitivity which will be measured using a 5-point ordinal scale (0=none, 1=minimal, 2=mild, 3=moderate, 4=severe).
Participant Assessment for Efficacy | Baseline, Week 2 and Week 4
  Participants observed efficacy parameters such as: smoothness, softness, clarity, radiance, pores and overall skin appearance which will be by using a 5-point ordinal scale (0=none, 1=minimal, 2=mild, 3=moderate, 4=severe).
Photographic Imaging (Right, Left and Frontal Face with Standard Lighting 1 and Cross Polarized Light) | Baseline, Week 2 and Week 4
  Photographic imaging (right, left and frontal face with standard lighting 1 and cross polarized light) will be obtained by using VISIA. Each participant's face will be imaged using the photographic imaging system prior to any product use. The imaging system takes a series of two high-resolution images that are captured sequentially in rapid succession to minimize panelist movement and maximize registration of images. Three sets of images will be taken - 45 degree left, 45 degree right, and center of the face.
Non-invasive Assessment: Transepidermal Water Loss (TEWL) | Baseline, Week 2 and Week 4
  TEWL measurements of defined target sites of face will be reported. A decrease in TEWL values reflects an improvement in the barrier properties of the skin.
Non-invasive Assessment: Skin pH | Baseline, Week 2 and Week 4
  Skin pH measurements of defined target sites of the face will be reported.
Non-invasive Assessment: Skin Hydration Measured by Corneometer | Baseline, Week 2 and Week 4
  Skin hydration of defined target sites of face as measured by Corneometer will be reported. An increase in values reflects an improvement in the hydration of the skin.
Non-invasive Assessment: Biomarker Tapes | Baseline, Week 2 and Week 4
  Three D-squame tape strips will be taken from a defined target site on the face. D-Squame Standard Sampling Discs (CuDerm Corporation, Dallas, N) will be used to non-invasively collect skin samples from the forehead. The discs are 2.2 centimeters (cm) in diameter and have a homogenous layer of a medical-grade adhesive, which safely removes stratum corneum components and provides optimum visibility of adhering corneocytes. Samples will be collected for the analysis of various skin biomarkers such as skin flakiness, as well as the integrity of the natural moisturizing factors (NMFs), ceramides, free fatty acids, cholesterol via biochemical assays.
Non-invasive Assessment: Facial Swabbing | Baseline, Week 2 and Week 4
  A swabbing technique will be used to collect surface skin microflora to determine the effect of the non-marketed cosmetic facial cleanser on the skin microflora.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Diana Draelos, MD, Principal Investigator — Dermatology Consulting Services, PLLC
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] U.S. Census Bureau. (n.d.). About race. Retrieved July 27, 2021, from https://www.census.gov/topics/population/race/about.html
- [Background] U.S. Census Bureau. (n.d.). About the Hispanic population and its origin. Retrieved July 27, 2021, from https://www.census.gov/topics/population/hispanic-origin/about.html
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKA004090&attachmentIdentifier=da2bc3db-39e3-4e8b-9c42-c66815e9ac6e&fileName=Summary_CSR_for_ClinTrials.gov_Posting.Pivotal.18NOV2022.pdf&versionIdentifier=